CLINICAL TRIAL: NCT06813612
Title: The Effects of Cognitive Behavioral Play Intervention on the Quality of Life of Children With Childhood-onset Epileptic Syndromes."
Brief Title: Effect of Cognitive Behavioral Play Intervention and Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Centro Ricerca "CBPT" Roma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: cbpt epi
Record Dates: First submitted 2025-01-10; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy; Epilepsy in Children
Keywords: epilepsy; psychology; cognitive behavioral play therapy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: patients consecutively enrolled will be assigned using a standard numerical randomization procedure. The randomization process will be carried out through the random sequence generator: www.randomizer.org. The required parameters will be entered into the generator (2 groups of 26 participants each for a sequence from 1 to 52 elements through extraction without replacement).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The person responsible for enrollment and the one responsible for pre- and post-intervention evaluations of participants will be blinded (single-blind) to the assignment to intervention conditions. Unblinding of the intervention condition may occur in the case of adverse clinical conditions that may arise during the study or due to the participants' early withdrawal from the study at their personal request.
  The person responsible for randomization and statistical analyses, as well as those who will administer the treatments, will be aware of the participants' assignment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition cognitive behavioral play intervention CBPI (Experimental): In the CBPI condition, children are given dolls and miniature props to play with, aiming to promote positive thinking. Each session includes stories on health, emotional well-being, social activities, and school life. The researcher teaches problem-solving by modeling steps like identifying the problem, generating solutions, evaluating them, and choosing the best solution. In each session, the researcher models the process four times and makes positive affirmations.
  The CBPI intervention and the free play control condition are similar, with both groups engaging in pretend play. The researcher uses standardized prompts and spends equal time and attention with each child. The key difference is that in the CBPI intervention, the researcher uses dolls to model positive thinking and problem-solving, while encouraging children's imagination and emotional expression. Techniques from play therapy are used to help children integrate their feelings into the stories
  Interventions: Behavioral: cognitive behavioral play intervention
- control condition of free playFP (No Intervention): The free play (FP) control condition allows the researcher to assess the effects of pretend play and provide positive attention to children. Children in this condition receive the same dolls and props, and hear the same stories as those in the cognitive-behavioral play intervention. After each story, they are encouraged to create their own story, but are free to play as they wish, often engaging in play unrelated to the story prompt. The researcher follows the child's lead, offering positive attention and non-specific praise but does not guide the play. The main difference between the two conditions is that in the FP condition, the researcher provides attention without directing the play, while in the intervention condition, the researcher actively guides the child's play to model problem-solving and positive thinking.

INTERVENTIONS:
Behavioral: cognitive behavioral play intervention — In the CBPI condition, children use dolls and miniature props to engage in play aimed at fostering positive thinking, a key element of quality of life. Each session includes stories on health, emotional well-being, social interactions, and school activities. The researcher demonstrates problem-solving steps, such as identifying and evaluating solutions, repeating this process three times. In each session, the researcher models problem-solving four times and provides at least five positive affirmations. Both the CBPI intervention and the free play control condition are similar, with the researcher using standardized prompts and providing equal time and positive attention. The key difference is that in the CBPI condition, the researcher models positive thinking and problem-solving, while in the free play condition, the researcher follows the child's lead without guiding play.
  Arms: Experimental condition cognitive behavioral play intervention CBPI

SUMMARY:
The goal of this clinical trial is to assess the effectiveness of Cognitive Behavioral Play Therapy interventions in patients with epilepsy.

Children with epilepsy will be randomly assigned to one of two intervention conditions: the experimental group will receive cognitive-behavioral play intervention, while the control group will engage in free play. Assessments will be done at the start (T0) and end (T1) of the intervention, measuring behaviors, coping strategies, positive thinking, problem-solving, and quality of life.

DETAILED DESCRIPTION:
Cognitive-Behavioral Play Therapy (CBPT) adapts Cognitive-Behavioral Therapy techniques into a play-based intervention for preschool and school-age children, especially for those facing challenges like hospitalization or chronic illnesses. Studies show that play has therapeutic value, helping children understand critical events, reduce anxiety, and cope with illness. This research aims to explore how CBPT can be applied in hospitals, specifically for children with epilepsy, to improve their quality of life, enhance problem-solving, and foster positive coping strategies. The goal is to validate CBPT as a supportive tool for enhancing psycho-emotional development and complementing medical care in hospital settings.

The study proposes a randomized controlled trial with two groups: children with epilepsy will be randomly assigned to either the cognitive-behavioral play intervention or free play. The study will assess internalizing and externalizing behaviors, coping strategies, positive thinking, problem-solving skills, and quality of life at baseline (T0) and after the 8 intervention sessions (T1).

The goal is to determine whether cognitive-behavioral play improves quality of life more than free play.

Both groups will participate in 8 weekly 40-minute play sessions, with an initial and final meeting to administer the questionnaires.

The psychologist conducting the assessments will be unaware of group assignments.

The play scenarios for both groups will be identical and based on common issues faced by children with epilepsy.

ELIGIBILITY:
For the purposes of the study, children aged between 6 and 10 years, of both sexes, will be recruited.

- inclusion criteria Children diagnosed with the following types of epilepsy will be included: childhood self-limiting focal epilepsy (SeLFE); childhood absence epilepsy (CAE); self-limiting centrotemporal paroxysmal epilepsy (SeLECTS); self-limiting epilepsy with autonomic seizures (SeLEAS); childhood occipital epilepsy (COVE); photosensitive occipital lobe epilepsy (POLE).

Exclusion criteria:

* Children with epilepsy in comorbidity with cognitive disabilities (the relevant cognitive disabilities must be specified with IQ scores)
* reduced visual or expressive hearing acuity (visually impaired or deaf) will be excluded.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
effect of cognitive behavioral play intervention on quality of life | 2 months
  To assess whether there is an improvement in the quality of life in children with epilepsy following a cognitive-behavioral play intervention , and whether these improvements are greater in this group compared to the control group.
  The Pediatric Quality of Life Inventory (PedsQL) Epilepsy Module will be used to measure the variable targeted by the intervention. The questionnaire uses a 5-point scale ranging from 0 (Never a problem) to 4 (Almost always a problem) for child and parent-report forms. For overall scores, it's possible to calculate a summary score with a range from 0 (worst possible health-related quality of life) to 100 (best possible health-related quality of life). Higher scores on the PedsQL Epilepsy Module indicate a better outcome, reflecting better health-related quality of life. Lower scores suggest a worse outcome.

SECONDARY OUTCOMES:
effect of cognitive behavioral play intervention on coping strategies | 2 months
  To verify whether a cognitive-behavioral play intervention, structured according to the theoretical framework of Cognitive Behavioral Play Therapy, can lead to an improvement in using standardized questionnaire The Children's Coping Strategies Checklist-Revised (CCSC-R1). The CCSC-R1 uses a Likert-type scale, typically ranging from 1 (Never use this strategy) to 5 (Always use this strategy) for each individual item. The total score depends on how the individual items are scored, but overall, higher scores represent greater use of coping strategies.
  Higher scores generally indicate greater use of coping strategies by the child. This is not necessarily a "better" or "worse" outcome in itself, but the effectiveness of coping strategies would depend on the context and type of coping used. For instance, adaptive coping strategies are generally considered positive, while maladaptive coping strategies might indicate poorer outcomes.
effect of cognitive behavioral play intervention on positive thinking | 2 months
  To verify whether a cognitive-behavioral play intervention, structured according to the theoretical framework of Cognitive Behavioral Play Therapy, can lead to an improvement in positive thinking,using standardized questionnaire: Positive Thinking Checklist (Checklist sul Pensiero Positivo) The scale typically uses a Likert-type scale ranging from 1 (Never) to 5 (Always), assessing how often an individual engages in positive thinking behaviors. Higher scores indicate more frequent use of positive thinking strategies, which generally reflect a better outcome, suggesting a more positive mindset or a greater tendency toward constructive thinking.

CONTACTS AND LOCATIONS:
Overall Officials: martina paola p zanaboni, psy, Principal Investigator — IRCCS Mondino Foundation
Locations (1):
- Child Neuropsichiatry, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Specchio N, Wirrell EC, Scheffer IE, Nabbout R, Riney K, Samia P, Guerreiro M, Gwer S, Zuberi SM, Wilmshurst JM, Yozawitz E, Pressler R, Hirsch E, Wiebe S, Cross HJ, Perucca E, Moshe SL, Tinuper P, Auvin S. International League Against Epilepsy classification and definition of epilepsy syndromes with onset in childhood: Position paper by the ILAE Task Force on Nosology and Definitions. Epilepsia. 2022 Jun;63(6):1398-1442. doi: 10.1111/epi.17241. Epub 2022 May 3. PMID 35503717